CLINICAL TRIAL: NCT04853420
Title: Minimal Residual Disease: A Trial Using Liquid Biopsies in Solid Malignancies.
Acronym: MARTINI
Status: Active, not recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0792
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-03

CONDITIONS: Cancer
Keywords: Minimal Residual Disease; liquid biopsy; ctDNA
MeSH Terms: conditions — Neoplasms; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The NHS' Genomic Medicine Service offers whole genome sequencing as part of the drive to improve cancer outcomes. It is recognised that actionable mutations (current and emerging), will ultimately improve outcomes across multiple disease sites by identifying which treatments may benefit individual patients the most, and by providing earlier and more accurate diagnoses. However, testing in the cancer setting is currently limited to haematological malignancies and sarcoma. The majority of patients with solid tumours do not yet have access to this platform and the benefits that it may bring. Therefore, expanding genomic testing capacity within a research setting has potential to benefit those patients that would otherwise not be able to access testing. In this study we will be using tissue derived from patients undergoing surgery for cancer to validate an in-house genomic testing platform against Roche's Foundation Medicine genomic profile service, which is an FDA- approved commercial platform.

In addition, two blood samples will be taken in order that we can test whether markers present in the tissue may also be seen in blood. We hope that this will help us monitor minimal residual disease in patients, allowing earlier detection of relapse/recurrence than radiology currently allows.

Patients may also agree to donate optional excess fresh tissue from their surgery. This will be integrated with other laboratory platforms which may offer information on prospective drug response based on genotypic profiles (e.g., patient-derived explants).

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Diagnosed with solid tumour that requires surgical resection, and has a high propensity of relapse.
* Fit for planned surgical procedure.
* Able (in the Investigators opinion) and willing to comply with all study requirements.
* Willing to allow his or her General Practitioner, Consultant, and Clinical Geneticist, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Female participants who are pregnant, lactating or planning pregnancy during the course of the study.
* Not fit for surgery.
* Not willing to donate blood and tissue samples.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Participants who have participated in another research study involving an investigational product in the past 12 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trial participants will consist of patients with solid tumours that have a high likelihood of rapid post-surgical relapse. Such tumours types typically include gastroesophageal, gastrointestinal cancers and colorectal liver metastases, but other malignancies will also be considered.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Cross-validate the in-house genetic testing platform against the FDA approved Foundation Medicine | 12-24 months
  To cross-validate the Thermofisher Oncomine tissue and cfTNA assays (in house) against the FDA approved Foundation Medicine platform by comparison of the spectrum and variant frequency of cancer-specific alterations detected in matched tissue and blood.

SECONDARY OUTCOMES:
Assess Utility in detecting minimal residual disease | 12-24 months
  To compare ctDNA mutations and variant frequency in blood samples pre- and post-surgery to assess utility in detection of minimal residual disease
Data integration | 12-24 months
  Ability to integrate data from clinical risk factors, and up-front genotyping.
Feasibility of testing platform in clinical setting | 12-24 months
  Feasibility of returning laboratory analysis in a clinically meaningful timeframe.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Thomas, Principal Investigator — University of Leicester/University Hospitals Leicester
Locations (1):
- University Hospitals of Leicester, Leicester, United Kingdom